CLINICAL TRIAL: NCT04496986
Title: Mechanisms, Predictors and Clinical Markers of Dysphagia in Cardiac Surgical Patients
Brief Title: Dysphagia in Cardiac Surgical Patients_
Status: Withdrawn | Type: Observational
Why Stopped: This study was replaced by a new study given recent funding by the NIH.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202001367; OCR39324 (Other: OCR OnCore)
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases
Keywords: Dysphagia; Extubation; Vocal Fold Mobility Impairment; Peak Cough Flow (PCF)
MeSH Terms: conditions — Cardiovascular Diseases; Deglutition Disorders | interventions — Pefloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiovascular Surgical Patients Preoperative Exam: All enrolled participants will undergo a baseline Fiberoptic Endoscopic Evaluation of Swallowing (FEES) before their surgery to determine baseline / preoperative swallowing function. Those with confirmed dysphagia will not be asked to complete the postoperative swallowing exam, given our desire to examine contributing risk factors for dysphagia development and mechanisms within cardiovascular surgical patients. In addition to the instrumental exam, systematic collection of demographic, medical, surgical, and intubation-related candidate predictor variables will be conducted over the entire perioperative period.
  Interventions: Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing
- Cardiovascular Surgical Patients Postoperative Exam: All remaining participants without preoperative dysphagia will be seen for a postoperative exam performed within 48 hours of extubation. Simultaneous imaging using FEES and videofluoroscopy will be performed at the bedside, as well as a battery of clinical tests. Completion of these postoperative tests will indicate study completion for participants without evidence of dysphagia, while participants who demonstrate acute-phase postoperative dysphagia will continue to participate if they desire. During their standard of care one-month follow-up appointment, a third research evaluation will be offered for participants with previously identified postoperative dysphagia. During this exam, the same imaging and clinical tests from the previous research exam will be performed. Finally, participants with persisting dysphagia will be offered the opportunity to continue to be studied for a fourth and final research exam during their standard of care six-month follow up clinic visit.
  Interventions: Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing; Diagnostic Test: Simultaneous FEES and Videofluoroscopy instrumental swallowing exam; Other: Voluntary Cough Peak Expiratory Flow (PEF) Testing; Other: Reflex Cough Screen; Other: Lingual Pressure Testing; Diagnostic Test: Speech Testing

INTERVENTIONS:
Diagnostic Test: Fiberoptic Endoscopic Evaluation of Swallowing — This procedure involves inserting a flexible laryngoscope that contains a light source and video camera on the end through the open passage of the nose towards the back of the throat in order to visualize the swallowing mechanism.
  Other Names: FEES
Diagnostic Test: Simultaneous FEES and Videofluoroscopy instrumental swallowing exam — This procedure involves inserting a flexible laryngoscope that contains a light source and video camera on the end through the open passage of the nose towards the back of the throat in order to visualize the swallowing mechanism. The participant will be asked to perform some voicing tasks, once completed, a videofluoroscopic swallowing exam will occur at the same time. This is like moving x-ray of the participant swallowing foods and liquids (barium).
  Other Names: Endofluoroscopy
  Groups: Cardiovascular Surgical Patients Postoperative Exam
Other: Voluntary Cough Peak Expiratory Flow (PEF) Testing — Cough PEF will be performed to index a participant's physiologic airway defense capacity and strength. Testing will occur with the participant seated upright at 90 degrees using an analog peak flow meter with a one-way expiratory valve that prevents a participant from breathing air in from the device to reduce contamination.
  Groups: Cardiovascular Surgical Patients Postoperative Exam
Other: Reflex Cough Screen — Participants will be seated upright and administered reflex cough testing via a disposable adult aerosol mask with an attached nebulizer that contains a solution to elicit a cough response.
  Groups: Cardiovascular Surgical Patients Postoperative Exam
Other: Lingual Pressure Testing — Lingual strength will be evaluated using the Iowa Oral Pressure Instrument (IOPI). Participants will be seated upright, and the SLP will place the IOPI air-filled sensing bulb in the midline anterior position on the participant's tongue, posterior to the alveolar ridge.
  Groups: Cardiovascular Surgical Patients Postoperative Exam
Diagnostic Test: Speech Testing — Speech assessment will occur with the participant comfortably seated headset microphone with a lapel windscreen connected to a TASCAM DR40 to allow for high-quality audio recordings. Individuals will be asked to perform two maximal performance speech tasks that include vowel prolongation of /a/, and a Diadochokinetic (DDK) rate task to examine SMR for production of the word "buttercup."
  Groups: Cardiovascular Surgical Patients Postoperative Exam

SUMMARY:
The proposed study seeks to determine the incidence of dysphagia and vocal fold mobility impairment (VFMI) in individuals undergoing cardiovascular surgical procedures. It also seeks to determine the impact of postoperative swallowing impairment on health-related outcomes.

DETAILED DESCRIPTION:
Swallowing impairment and VFMI are common, yet often overlooked, complications of cardiovascular surgical procedures. The true incidence of both dysphagia and VFMI in this patient population is unclear due to a lack of rigorous study using instrumental assessment techniques and validated outcomes in all patients undergoing cardiovascular surgery. The study is therefore aimed to determine the incidence of dysphagia and VFMI in this patient population and to characterize impairment profiles related to swallowing safety and efficiency. In addition, the study is also aimed to assess the relative impact of VFMI and dysphagia on health-related outcomes such as length of hospital stay, pneumonia, sepsis, reintubation, and discharge status. We will identify risk factors for postoperative dysphagia and VFMI in cardiovascular patients to build a practical electronic risk-stratification tool. We also aim to identify sensitive bedside clinical markers of dysphagia in postoperative cardiovascular patients to develop a bedside screening tool. All participants will undergo two research visits (one preoperatively and one postoperatively) where they will undergo an instrumental swallowing test and complete several patient report outcomes and clinical tests. If they are found to have dysphagia after surgery, they will be offered no-cost follow up swallow tests at months 1 and 6. Finally, health-related outcomes will be indexed in enrolled participants to determine the impact of dysphagia.

ELIGIBILITY:
Inclusion Criteria: 1) individuals over 18 years of age, 2) undergoing a cardiovascular procedure at the University of Florida Heart and Vascular Hospital, 3) confirmed negative COVID-19 test result, 4) no allergies to barium, 5) not pregnant (female participants), and 6) willing to participate in research exams.

Exclusion Criteria: 1) individuals under the age of 18, 2) patients with a confirmed positive COVID-19 test result, 3) participants with allergies to barium, 4) pregnant women, or 5) unwilling to participate in research exams.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 360 individuals undergoing cardiac surgery will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | Baseline (Prior to surgery)
  This scale is a validated measure used by trained blinded clinicians to assign ratings of safety to swallowing bolus trials. The development and use of an 8-point, equal-appearing interval scale (8 being best; 1 being worst) to describe penetration and aspiration events are described. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled. (FEES)
Penetration Aspiration Scale | Follow-up - Within 72 hours following extubation from surgery and onward
  This scale is a validated measure used by trained blinded clinicians to assign ratings of safety to swallowing bolus trials. The development and use of an 8-point, equal-appearing interval scale (8 being best; 1 being worst) to describe penetration and aspiration events are described. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled. (Used in both FEES and VFSS)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Plowman, PhD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No